CLINICAL TRIAL: NCT07050524
Title: Evaluating the Effect of Omega-3 Fatty Acids Supplementation on the Efficacy of Neoadjuvant Immunotherapy in Patients With Locally Advanced Gastric and Gastroesophageal Junction Adenocarcinoma: A Multicenter, Randomized, Controlled Phase II Clinical Trial
Brief Title: Omega-3 Supplementation and Immunotherapy in Gastric Cancer: A Phase II Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Affiliated Jiangning Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSIRIS
Record Dates: First submitted 2025-06-26; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer Stage III
Keywords: omega-3; Neoadjuvant Immunotherapy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This interventional study employs a randomized, controlled design to evaluate the effects of Omega-3 fatty acids supplementation on the efficacy of neoadjuvant immunotherapy in patients with locally advanced gastric and gastroesophageal junction adenocarcinoma. Participants will be randomly assigned to one of two groups: the experimental group receiving Omega-3 supplementation alongside standard neoadjuvant immunotherapy, and the control group receiving only the standard immunotherapy. The primary endpoints include pathologic complete response (pCR) rates and major pathological response (MPR) rates. The study will also assess secondary outcomes such as nutritional status, immune function, inflammatory responses, adverse events, and quality of life metrics. By utilizing a controlled framework, this study aims to provide robust evidence regarding the potential benefits of Omega-3 supplementation in enhancing immunotherapy outcomes for gastrointestinal cancers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Receiving Omega-3 supplementation alongside standard neoadjuvant immunotherapy
  Interventions: Dietary Supplement: Omega-3 Supplementation; Drug: Neoadjuvant Immunotherapy
- control group (Active Comparator): Receiving only the standard immunotherapy
  Interventions: Drug: Neoadjuvant Immunotherapy

INTERVENTIONS:
Dietary Supplement: Omega-3 Supplementation — Participants assigned to the experimental group will receive Omega-3 fatty acids supplementation as part of their treatment regimen. The Omega-3 supplementation will consist of high-quality fish oil capsules, providing a daily dose of [specific dosage, e.g., 2000 mg of EPA and DHA combined], taken orally. This supplementation will commence concurrently with the initiation of neoadjuvant immunotherapy and will continue throughout the treatment period.
  Arms: experimental group
Drug: Neoadjuvant Immunotherapy — Participants in both the experimental and control groups will receive neoadjuvant immunotherapy designed to stimulate the body's immune response against locally advanced gastric and gastroesophageal junction adenocarcinomas. The specific regimen will involve administration of [specific immunotherapeutic agents, e.g., pembrolizumab, nivolumab, etc.] in accordance with established clinical protocols.
  The neoadjuvant immunotherapy will be administered through intravenous infusion, typically starting [specify timeline, e.g., 4-6 weeks] prior to surgical resection of the tumor. Treatment cycles will be scheduled every [specify interval, e.g., 2 or 3 weeks], depending on the specific agent used and participant response.

SUMMARY:
The goal of this clinical trial is to learn if Omega-3 fatty acids supplementation can enhance the efficacy of neoadjuvant immunotherapy in patients with locally advanced gastric and gastroesophageal junction adenocarcinoma. The main questions it aims to answer are: does Omega-3 supplementation improve the pathologic complete response (pCR) rate compared to standard neoadjuvant immunotherapy alone, and is there an increase in the major pathological response (MPR) rate with Omega-3 supplementation? Researchers will compare the group receiving Omega-3 supplementation with the control group receiving standard neoadjuvant immunotherapy to see if Omega-3 supplementation leads to better treatment outcomes. Participants will receive Omega-3 fatty acids supplements in conjunction with their prescribed neoadjuvant immunotherapy, undergo regular assessments of their pathologic response to treatment, and provide information on their nutritional status and quality of life throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Participants must be aged 18 years or older.
2. Diagnosis: Confirmed diagnosis of locally advanced gastric or gastroesophageal junction adenocarcinoma, classified as clinical stage II or III according to the American Joint Committee on Cancer (AJCC) staging system.
3. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, indicating that patients are fully active or restricted in physically strenuous activity but are capable of self-care.
4. Histological Verification: Tissue confirmation of diagnosis must be obtained via biopsy, with adequate archival tumor tissue available for biomarker analysis if required.
5. Organ Function: Adequate organ function as evidenced by laboratory tests:

   Absolute neutrophil count (ANC) ≥ 1,500/mm³ Platelet count ≥ 100,000/mm³ Hemoglobin ≥ 9 g/dL Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) Total bilirubin ≤ 1.5 times the ULN (unless due to Gilbert's syndrome) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the ULN (≤ 5 times the ULN if liver metastases are present)
6. Informed Consent: Ability and willingness to provide written informed consent prior to any study-related procedures.

Exclusion Criteria:

1. Previous Therapy: Prior treatment with chemotherapy, radiation therapy, or immunotherapy for the current cancer diagnosis.
2. Concurrent Malignancies: Presence of another active malignancy within the past 5 years (except for non-melanoma skin cancer or cervical carcinoma in situ).
3. Active Infection: Presence of any uncontrolled infection requiring systemic therapy or serious co-morbid conditions that would compromise program compliance or interfere with study results.
4. Allergies: Known hypersensitivity or contraindications to Omega-3 fatty acid supplementation or components of the immunotherapy regimen.
5. Pregnancy/Breastfeeding: Women who are pregnant or breastfeeding; fertile men and women not employing effective contraception during the study period.

Psychiatric Condition: Any psychiatric condition or substance abuse that would interfere with compliance or affect the participant's safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | 8 to 12 weeks

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | 8 to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China